CLINICAL TRIAL: NCT01738880
Title: Effect of Goal-directed Fluid Therapy Based on Stroke Volume Variation on Metabolic Acidosis in Patients Undergoing Brain Tumor Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2012-0404
Record Dates: First submitted 2012-11-18; First posted 2012-11-30 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group C (Active Comparator): intraoperative fluid management based on CVP
  Interventions: Drug: CVP
- group S (Experimental): intraoperative fluid management based on SVV
  Interventions: Drug: SVV

INTERVENTIONS:
Drug: SVV — During the surgery, patients in group S receive additional fluids (400 ml of normal saline or 200 ml of colloid) when SVV is less than 13.
  Arms: group S
Drug: CVP — Patients in group C receive additional fluids (400 ml of normal saline or 200 ml of colloid) when CVP is less 8 during the surgery.
  Arms: group C

SUMMARY:
In patients undergoing craniotomy, 0.9% normal saline is commonly administered in order to reduce cerebral edema. Excessive administration of 0.9% normal saline has been to reported to cause hyperchloremic metabolic acidosis. On the other hand, hypovolemia due to insufficient fluid replacement for perioperative loss can also result in metabolic acidosis by lactic acid accumulation. However, the guideline for perioperative fluid management has not been yet established. The investigators hypothesized that intraoperative fluid management according to SVV(Stroke Volume Variation)could reduce perioperative metabolic acidosis compared to those by CVP(Central Venous Pressure). Therefore, the study is trying to determine if intraoperative fluid administration based on SVV could reduce metabolic acidosis when compared with CVP in patients undergoing craniotomy due to brain tumor who receive 0.9% normal saline as main fluid regimen.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing craniotomy due to brain tumor
* American Society of Anesthesiologists physical status I or II
* aged from 20 to 65

Exclusion Criteria:

* compromised cardiopulmonary function
* diabetes mellitus
* symptom or sign with increased intracranial pressure
* liver or renal disease
* pre-existing metabolic acidosis
* pregnant or breast-feeding
* patients who cannot understand the statements for subjects

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Standard base excess point | at the suturing of scalp

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea